CLINICAL TRIAL: NCT06739824
Title: Comparison of Spencer Technique and Conventional Treatment in Adjuncts to Corticosteroid Injection in Frozen Shoulder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/762
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Frozen Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental)
  Interventions: Diagnostic Test: Conventional Treatment(CI)
- EXP group (Active Comparator)
  Interventions: Combination Product: Spencer Technique (CI)

INTERVENTIONS:
Diagnostic Test: Conventional Treatment(CI) — Patients receive a corticosteroid injection followed by conventional treatment, such as standard physical therapy exercises focused on range of motion and strengthening, without the specific manual techniques of the Spencer method.
  Arms: Control Group
Combination Product: Spencer Technique (CI) — Patients receive a corticosteroid injection followed by the Spencer technique, which involves a series of specific manual mobilization maneuvers aimed at improving shoulder mobility and reducing pain.
  Arms: EXP group

SUMMARY:
This study will compare the effectiveness of the Spencer Technique combined with intra-articular injection versus conventional therapy combined with intra-articular injection in managing frozen shoulder. The research problem addresses the need for optimal therapeutic approaches to improve pain relief, range of motion, and functional recovery in patients with frozen shoulder.

DETAILED DESCRIPTION:
Utilizing a randomized controlled trial, the study will recruit 100 participants, divided into two groups: Group A receiving the Spencer Technique with intra-articular injection and Group B receiving conventional therapy with intra-articular injection. Outcome measures will include pain levels, range of motion, shoulder functional status and patient satisfaction, assessed through validated tools. The significance of this study lies in its potential to provide robust comparative data to guide clinical decisions and enhance patient outcomes, particularly in populations with a high prevalence of diabetes

ELIGIBILITY:
Inclusion Criteria:

* 30 years 60 years old.
* Diagnosed with unilateral adhesive capsulitis presenting symptoms of pain.
* restricted range of motion of frozen shoulder Stage 2 and 3

Exclusion Criteria:

* Rotator cuff injury
* Long-term Systemic Corticosteroid use
* Previous Ipsilateral shoulder CSI within 12 months.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Functional Shoulder Scale | 12 Months
  This tool includes a pain scale with a score of 1 to 10 and daily activity scales, including 10 activities. Each activity has a score of 1 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- New Haider Hospital/THQ Muridke, Sheikhupura, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No